CLINICAL TRIAL: NCT06156332
Title: A Single-arm, Single-center, Phase II Clinical Study of Surufatinib Combined With Serplulimab in the Treatment of Advanced Solid Tumors With Neuroendocrine Differentiation That Failed Standard Therapy
Brief Title: A Study of Surufatinib Combined With Serplulimab in the Treatment of Advanced Solid Tumors With Neuroendocrine Differentiation That Failed Standard Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Oncology department chief physician, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFSL-NED
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors With Neuroendocrine Differentiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surufatinib combined with serplulimab (Experimental): surufatinib: 250 mg (5 capsules) once a day, Q3W, continued until the patient developed disease progression or met other protocol criteria for discontinuation of study treatment; If the patient vomits after taking the medicine, there is no need to take the supplement; The missed dose should not be added the next day, and the next prescribed dose should be taken as usual.
  serplulimab: 300mg fixed dose, intravenous infusion, d1, Q3W; Continued administration until the patient developed disease progression or met other protocol criteria for discontinuation of study therapy.
  Interventions: Drug: surufatinib、serplulimab

INTERVENTIONS:
Drug: surufatinib、serplulimab — surufatinib:
  250 mg (5 capsules) once a day, Q3W, continued until the patient developed disease progression or met other protocol criteria for discontinuation of study treatment; If the patient vomits after taking the medicine, there is no need to take the supplement; The missed dose should not be added the next day, and the next prescribed dose should be taken as usual.
  serplulimab:
  300mg fixed dose, intravenous infusion, d1, Q3W; Continued administration until the patient developed disease progression or met other protocol criteria for discontinuation of study therapy.
  Imaging was used every 6 weeks (±7 days) to evaluate tumor status until disease progression (RECIST 1.1) or death (during patient treatment), and tumor treatment and survival status after disease progression were recorded. The changes of neuroendocrine tumor markers were detected after treatment.

SUMMARY:
Enrolled patients with advanced solid tumors with neuroendocrine differentiation who had failed standard therapy (including those with initial advanced solid tumors with neuroendocrine differentiation and those with newly developed neuroendocrine differentiation after treatment failure) received the combination of serplulimab and surufatinib and continued to be administered until the patient developed disease progression or met other protocol criteria for discontinuation of study therapy. A total of 39 patients were enrolled.

ELIGIBILITY:
Inclusion Criteria:

-

1. Age ≥18 years old;

2. Histologically confirmed locally advanced late or metastatic unresectable solid tumors (lung cancer, gastric cancer, bowel cancer, etc.) with NED (neuroendocrinization, positive expression of at least one neuroendocrine marker CgA or Syn by immunohistochemistry), the initial standard treatment response is significantly lower than expected (tumor regression is not obvious, or PFS duration is short, as determined by the investigator);

1. Lung cancer: Locally advanced or metastatic (stage IIIB, IIIC, or IV) non-squamous non-small cell lung cancer (NSCLC) that is histologically or cytologically confirmed to be inoperable and not subject to radical concurrent radiotherapy and chemotherapy (according to the AJCC staging system Edition 8); Based on tissue examination, EGFR sensitive mutation, ALK, ROS1 gene fusion mutation was not detected driver gene negative;
2. Gastric cancer: histologically or pathologically confirmed advanced HER-2 negative gastric adenocarcinoma (including adenocarcinoma of the gastroesophageal junction);
3. Colorectal cancer: On the basis of adenocarcinoma diagnosis of colorectal cancer, morphologic neuroendocrine differentiation phenotype appears;
4. Breast cancer: histologically or pathologically confirmed advanced breast cancer, HER-2 negative;
5. Prostate cancer: advanced prostate cancer confirmed by histology or pathology, with positive staining of specific markers;

3.ECOG score: 0-1;

4. Patients with advanced solid tumors (lung cancer, stomach cancer, bowel cancer, etc.) with new neuroendocrine differentiation after previous standard treatment failure (or intolerance);

5. There is at least one CT measurable lesion according to RECIST 1.1 criteria;

6. Expect to survive for at least 3 months.

(7) Patients of reproductive age (including female and male patients' female companions) must use effective birth control measures;

8. Subjects voluntarily join the study and sign an informed consent form (ICF);

9. It is expected that the compliance is good, and the efficacy and adverse reactions can be followed up according to the protocol requirements.

Exclusion Criteria:

1. Received the following treatments within 4 weeks of treatment: including but not limited to surgery, chemotherapy, radical radiotherapy, biological targeted therapy, immunotherapy, anti-tumor Chinese medicine therapy, interventional embolization of hepatic artery, liver metastasis cryoablation or radiofrequency ablation of tumor radiation therapy, and other clinical investigational drugs;
2. Patients who have previously used surufatinib and or Srulizumab
3. Pregnant or lactating women;
4. Patients who have participated in other clinical trials and have not yet terminated the trial;
5. Patients with a definite tendency to gastrointestinal bleeding. Including the following conditions: ① there are locally active ulcer lesions, and stool occult blood 2+ or more; (Fecal occult blood 2+ was allowed to re-test fecal occult blood, and patients who were judged by the investigator to have clear benefits could be enrolled); ② Patients with history of black stool and hematemesis within 3 months;
6. Major organ functions within 7 days prior to treatment meet the following criteria:

(1) Hemoglobin (HB) ≤90 g/L;

(2) Absolute value of neutrophil (ANC) ≤1.5×109/L;

(3) Platelet (PLT) ≤100×109/L.

7. Biochemical examination shall meet the following standards:

1. Total bilirubin (TBIL) ≥1.5 times the upper limit of normal (ULN);
2. Alanine aminotransferase (ALT) and aspartate aminotransferase AST≥2.5×ULN, if accompanied by liver metastasis, ALT and AST≥5×ULN;
3. Serum creatinine (Cr) ≥1.5×ULN or creatinine clearance (CCr)≤60ml/min;

8. Patients with any severe and/or uncontrolled disease, including:

1. Patients with unsatisfactory blood pressure control (systolic pressure ≥150 mmHg, diastolic pressure ≥100 mmHg);
2. have grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480ms), and ≥ grade 2 congestive heart failure (NYHA);
3. Active or uncontrolled severe infection (≥CTC AE grade 2 infection);
4. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy;
5. Renal failure requires hemodialysis or peritoneal dialysis;
6. Two consecutive urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0 g;
7. Suffering from mental illness, including epilepsy, dementia, severe depression, mania, etc.

9. Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to the grouping (specifically in conjunction with clinical evaluation);

10. With pleural effusion or ascites, causing respiratory syndrome (≥CTC AE grade 2 dyspnea);

11. Patients who had received chemotherapy, radiotherapy, or other experimental anti-cancer treatment (other than bisphosphonate) within 4 weeks prior to the first dosing of this study. Those who had previously received local radiotherapy were eligible if they met the following criteria: more than 4 weeks from the end of radiotherapy to the start of the study (more than 2 weeks for brain radiotherapy); In addition, the target lesions selected in this study were not in the radiotherapy area, or if the target lesions were in the radiotherapy area but had confirmed progression;

12. History of any active autoimmune disease or autoimmune disease, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, pituitary inflammation, vasculitis, systemic lupus erythematosus, etc.;

13. Patients whose imaging shows that the tumor has invaded important blood vessels, or who are judged by the investigators to be highly likely to invade important blood vessels and cause fatal major bleeding during follow-up studies;

14. Patients with any physical signs or history of bleeding, regardless of severity; Patients with any bleeding or bleeding events ≥CTCAE grade 3, unhealed wounds, ulcers, or fractures during the first 4 weeks of enrollment;

15. Have a history of other malignant tumors within five years, except for cured cervical carcinoma in situ or skin basal cell carcinoma;

16. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;

17. Patients with severe allergic history or allergic constitution;

18. Patients with brain metastases accompanied by symptoms or symptoms controlled for less than 2 months;

19. Any disease or condition affecting the absorption of the drug, or inability to take the investigational drug orally;

20. The researcher considers that there are other circumstances that are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-28 (Estimated); Primary Completion 2025-01-28 (Estimated); Study Completion 2027-01-28 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of enrollment until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Objective response rate

SECONDARY OUTCOMES:
PFS | From date of randomization until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival
OS | From date of randomization until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Overall survival
DCR | From date of randomization until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Sheng Zang, Principal Investigator — Shanghai Changzheng Hospital

IPD SHARING:
Plan to Share IPD: No